CLINICAL TRIAL: NCT04922866
Title: Predictive Nomogram for Postoperative Acute Kidney Injury (AKI) in Elderly Patients Following Liver Resection
Status: Completed | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Weidong Mi, Director (Cheif expert of National key research and development program of China 2018YFC2001900), Chinese PLA General Hospital
Other Study IDs: PLAGH-AOC-002
Record Dates: First submitted 2021-06-07; First posted 2021-06-11 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Postoperative Acute Kidney Injury
Keywords: acute kidney injury; predictive nomogram; elderly; liver resection
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- elderly patients following hepatectomy: elderly patients (aged ≥65 years) scheduled for any type of liver resection
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Acute kidney injury (AKI) is a severe complication after liver resection and is associated with morbidity and mortality. The incidence of postoperative AKI is significantly higher in elderly patients, especially in those with comorbidities.

There is currently limited evidence on the incidence and associations of postoperative AKI in elderly patients following liver resection.

This study will evaluate the incidence and associations of AKI in elderly patients after liver resection and its impact on postoperative mortality.

DETAILED DESCRIPTION:
The occurrence of postoperative AKI is independently associated with increased morbidity and mortality. Advanced age reduces renal autoregulatory capacity due to physiological and functional changes, thus render the elderly to suffer postoperative AKI and probably the consequent chronic kidney disease.

Although elderly patients account for approximately 25% of surgical procedures, the incidence and associations of AKI in this group of patients are rarely understood.

Thus, it is essential to identify those patients at high risk to develop postoperative AKI to optimize perioperative prevention and protection strategies.

This study is a retrospective cohort study, aim to access risk factors of postoperative AKI and its association with outcomes. The investigators will develop and validate a predictive model for postoperative AKI.

The principal clinical outcome of the study is postoperative AKI, defined as an absolute increase in serum creatinine of 0.3 mg/dL within 48 hours or a 1.5-fold increase from preoperative baseline within seven days after surgery, according to the Kidney Disease: Improving Global Outcomes (KDIGO) criterion.

ELIGIBILITY:
Inclusion Criteria:

* Elderly patients aged ≥65 years
* Benign and malignant liver diseases

Exclusion Criteria:

* Emergency operation
* Liver transplantation

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly patients (aged ≥ 65 years) with benign and malignant liver diseases of the Chinese PLA General Hospital HPB (Hepato-Pancreato-Biliary) Center undergoing liver resection from 2012-2019
Sampling Method: Non-Probability Sample
Enrollment: 843 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Postoperative acute kidney injury | postoperative seven days
  Postoperative acute kidney injury is defined as an absolute increase in serum creatinine of 0.3 mg/dl within 48 hours or a 1.5-fold increase from preoperative baseline within seven days after surgery, according to the Kidney Disease: Improving Global Outcomes (KDIGO) criterion.

SECONDARY OUTCOMES:
Incidence of postoperative AKI | postoperative seven days
  collection of clinical data in the medical record and follow-up update

CONTACTS AND LOCATIONS:
Overall Officials: Weidong Mi, PhD, Study Director — Chinese PLA General Hospital
Locations (2):
- China (2):
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Chinese PLA General Hospital, Beijing

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yu Y, Zhang C, Zhang F, Liu C, Li H, Lou J, Xu Z, Liu Y, Cao J, Mi W. Development and validation of a risk nomogram for postoperative acute kidney injury in older patients undergoing liver resection: a pilot study. BMC Anesthesiol. 2022 Jan 13;22(1):22. doi: 10.1186/s12871-022-01566-z. PMID 35026992